CLINICAL TRIAL: NCT05921331
Title: Mobile Medical Application on Adjuvant Therapy Compliance and Quality of Life in Patients With Early Breast Cancer: a Multicentric, Open-labeled, Randomized Controlled Trial
Brief Title: RJBC-APP and Breast Cancer Treatment Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RJBC-APP
Record Dates: First submitted 2023-05-02; First posted 2023-06-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The RJBC-APP group (Experimental): Participants randomized to the RJBC-APP group should register on the RJBC-APP, through which they can receive treatment reminders, matters needing attention as well as science knowledge and communicate with the medical staff.
  Interventions: Device: The RJBC-APP; Other: Routine post-surgical follow-up
- The Control group (Active Comparator): Participants randomized to the Control group have no access to the RJBC-APP and post-surgical follow-up can only be conducted in outpatient clinic.
  Interventions: Other: Routine post-surgical follow-up

INTERVENTIONS:
Device: The RJBC-APP — The RJBC-APP consists of the following features: 1. Login, logout, setting, and modification of personal information. 2. Full-course management included registering for information on the surgical treatment, viewing the results of the multidisciplinary team (MDT) discussion, generating the treatment process according to the MDT discussion, receiving the reminder of the treatment, confirming the completion of the treatment, filling in the follow-up information, and consulting a specialist nurse. 3. Questionnaire and feedback.
  Other Names: RJBC Full-Course Management APP
  Arms: The RJBC-APP group
Other: Routine post-surgical follow-up — The routine post-surgical follow-up is conducted in the outpatient clinic.

SUMMARY:
The goal of this multicentric randomized controlled clinical trial is to test the role of mobile medical application (APP) on adjuvant therapy compliance and quality of life (QoL) in patients with early breast cancer. Participants assigned to the Ruijin Breast Cancer APP (RJBC-APP) group can receive treatment reminders, matters needing attention as well as science knowledge and they can communicate with the medical staff during adjuvant treatments while follow-up can only be conducted in outpatient clinic for those in the Control group.

DETAILED DESCRIPTION:
Adjuvant treatments has significantly improved the prognosis of early breast cancer patients. However, previous studies suggested the existence of noncompliance to adjuvant therapies, which might cause detriments to disease outcomes. The goal of this multicentric randomized controlled clinical trial is to test the role of mobile medical application (APP) on adjuvant therapy compliance and quality of life (QoL) in patients with early breast cancer. Patients diagnosed with invasive breast cancers after surgery will be randomly assigned to the Ruijin Breast Cancer APP (RJBC-APP) group or the Control group. Those in the RJBC-APP group can receive treatment reminders, matters needing attention as well as science knowledge and they can communicate with the medical staff during adjuvant treatments while follow-up can only be conducted in outpatient clinic for those in the Control group. The primary endpoint is the rate of adjuvant therapy compliance at 12 months after randomization. Secondary endpoints consist of compliance rates at 3, 6, 24 months after randomization, QoL and cancer-related symptoms scores at 3, 6, 12, 24 months, disease-free survival (DFS) and overall survival (OS) at 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-70
2. Eastern Cooperative Oncology Group Performance Status Score 0-2
3. Breast cancer by pathology
4. Adjuvant therapy by multidisciplinary team
5. Written informed consent form

Exclusion Criteria:

1. Distant metastases at diagnosis
2. Unable to use a smartphone

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Rate of compliance with adjuvant therapy | 12 months after adjuvant therapy
  Compliance is defined as completing the adjuvant therapy recommended by multidisciplinary team in terms of the type, dosage, date and course, and non-compliance is considered in the presence of any of the following cases: 1) the patient refuses to accept the recommended treatments, 2) the actual treatments are different from those recommended, 3) the patient dose not complete the full course of treatments, 4) the patient starts the treatment 7 days or more later than the established date, 5) the patient does not follow the recommended dose and intensity.
Overall Survival (OS) | 60 months after adjuvant therapy
  OS is calculated from the date of surgery to the date of death.

SECONDARY OUTCOMES:
Rate of compliance with adjuvant therapy | 3、6 and 24 months after adjuvant therapy
  Compliance is defined as completing the adjuvant therapy recommended by multidisciplinary team in terms of the type, dosage, date and course, and non-compliance is considered in the presence of any of the following cases: 1) the patient refuses to accept the recommended treatments, 2) the actual treatments are different from those recommended, 3) the patient dose not complete the full course of treatments, 4) the patient starts the treatment 7 days or more later than the established date, 5) the patient does not follow the recommended dose and intensity.
Quality of Life (QoL) Scale | 3、6、12 and 24 months after adjuvant therapy
  The QoL Scale is evaluated by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30, version 3.0). The questionnaire is composed of 30 items among which items 1-28 are divided into 4 levels (scored as 1-4 respectively, higher scores mean a worse outcome) and items 29-30 are divided into 7 grades (scored as 1-7 respectively, higher scores mean a better score). The items are further divided into 15 domains. The standard score (0-100) is calculated from raw score of each domain and higher scores mean a better outcome.
Cancer-related symptoms scores | 3、6、12 and 24 months after adjuvant therapy
  Cancer-related symptoms are evaluated by the MD Anderson Symptom Inventory (MDASI). The questionnaire is composed of 19 items among which items 1-13 are degree of 13 common symptoms and items 14-19 are degrees of the impact on daily life (scored as 1-10 respectively, higher scores mean a better score). The total score (0-190) is calculated by sum of each item and higher scores mean a worse outcome.
Disease-free Survival (DFS) | 60 months after adjuvant therapy
  DFS is calculated from the date of surgery to the first date of the following events: local recurrence, regional recurrence, distant metastasis, contralateral breast cancer, secondary primary malignancy and death.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosong Chen, Professor, Principal Investigator — Xiaosong Chen
Locations (1):
- Xiaosong Chen, Shanghai, Please Select, China

IPD SHARING:
Plan to Share IPD: No